CLINICAL TRIAL: NCT01553591
Title: A Randomized, Double-blind, Placebo-controlled, Phase 3 Study to Evaluate the Efficacy, Safety, and Tolerability of JNJ-27018966 in the Treatment of Patients With Diarrhea-Predominant Irritable Bowel Syndrome
Brief Title: Efficacy, Safety, and Tolerability of Eluxadoline in the Treatment of Participants With Diarrhea-Predominant Irritable Bowel Syndrome (IBS-d)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Furiex Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 27018966IBS3001; 2012-001600-38 (EudraCT Number)
Record Dates: First submitted 2012-03-08; First posted 2012-03-14 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — eluxadoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Eluxadoline 75 mg (Experimental): Eluxadoline 75 mg tablets, orally, twice daily for up to 52 weeks period.
  Interventions: Drug: Eluxadoline
- Eluxadoline 100 mg (Experimental): Eluxadoline 100 mg tablets, orally, twice daily for up to 52 weeks period.
  Interventions: Drug: Eluxadoline
- Placebo (Placebo Comparator): Eluxadoline placebo matching tablets, orally, twice daily for up to 52 weeks period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eluxadoline — Oral tablets twice daily
  Other Names: JNJ-27018966
  Arms: Eluxadoline 100 mg; Eluxadoline 75 mg
Drug: Placebo — Oral tablets twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy, safety, and tolerability of different doses of eluxadoline (JNJ-27018966) compared with placebo in the treatment of participants with diarrhea-predominant irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has a diagnosis of irritable bowel syndrome (IBS) with a subtype of diarrhea defined by the Rome III criteria.
2. Participant has had a colonoscopy performed:

   * Within 10 years prior to Prescreening if participant is at least 50 years of age (sigmoidoscopy, double contrast barium enema, or computed tomography (CT) colonography within the past 5 years is acceptable)
   * Since the onset (if applicable) of any of the following alarm features for participants of any age:

     * Participant has documented weight loss within the past 6 months
     * Participant has nocturnal symptoms
     * Participant has a familial history of first-degree relatives with colon cancer or
     * Participant has blood mixed with their stool (excluding blood from hemorrhoids).
3. Female participants must be:

   * Postmenopausal, defined as 52 years or older and amenorrheic for at least 2 years at Prescreening,
   * Surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy),
   * Abstinent, or
   * If sexually active, be practicing an effective method of birth control.

Exclusion Criteria:

1. Participant has a diagnosis of IBS with a subtype of constipation, mixed IBS, or unsubtyped IBS by the Rome III criteria.
2. Participant has a history of inflammatory or immune-mediated gastrointestinal (GI) disorders including inflammatory bowel disease (ie, Crohn's disease, ulcerative colitis) and celiac disease.
3. Participant has a history of diverticulitis within 3 months prior to Prescreening.
4. Participant has a history of intestinal obstruction, stricture, toxic megacolon, GI perforation, fecal impaction, gastric banding, bariatric surgery, adhesions, ischemic colitis, or impaired intestinal circulation (eg, aortoiliac disease).
5. Participant has any of the following surgical history:

   * Cholecystectomy with any history of post cholecystectomy biliary tract pain
   * Any abdominal surgery within the 3 months prior to Prescreening
   * Participant has a history of major gastric, hepatic, pancreatic, or intestinal surgery (appendectomy, hemorrhoidectomy, or polypectomy greater than 3 months post surgery are allowed)

Other protocol-specific eligibility criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1282 (Actual)
Dates: Start 2012-05-29 (Actual); Primary Completion 2014-07-29 (Actual); Study Completion 2014-07-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (243):
- United States (218):
  - Furiex Research Site, Athens, Alabama
  - Furiex Research Site, Birmingham, Alabama
  - Furiex Research Site, Foley, Alabama
  - Furiex Research Site, Huntsville, Alabama
  - Furiex Research Site, Ozark, Alabama
  - Furiex Research Site, Chandler, Arizona
  - Furiex Research Site, Glendale, Arizona
  - Furiex Research Site, Mesa, Arizona
  - Furiex Research Site, Phoenix, Arizona
  - Furiex Research Site, Tucson, Arizona
  - Furiex Research Site, Little Rock, Arkansas
  - Furiex Research Site, North Little Rock, Arkansas
  - Furiex Research Site, Azusa, California
  - Furiex Research Site, Bell Gardens, California
  - Furiex Research Site, Beverly Hills, California
  - Furiex Research Site, Carson, California
  - Furiex Research Site, Chula Vista, California
  - Furiex Research Site, Corona, California
  - Furiex Research Site, El Cajon, California
  - Furiex Research Site, Encino, California
  - Furiex Research Site, Garden Grove, California
  - Furiex Research Site, Lomita, California
  - Furiex Research Site, Los Angeles, California
  - Furiex Research Site, Monterey Park, California
  - Furiex Research Site, Murrieta, California
  - Furiex Research Site, Newport Beach, California
  - Furiex Research Site, North Hollywood, California
  - Furiex Research Site, Oakland, California
  - Furiex Research Site, Oxnard, California
  - Furiex Research Site, Pismo Beach, California
  - Furiex Research Site, Poway, California
  - Furiex Research Site, Riverside, California
  - Furiex Research Site, Roseville, California
  - Furiex Research Site, Sacramento, California
  - Furiex Research Site, San Diego, California
  - Furiex Research Site, Santa Monica, California
  - Furiex Research Site, Thousand Oaks, California
  - Furiex Research Site, Colorado Springs, Colorado
  - Furiex Research Site, Lafayette, Colorado
  - Furiex Research Site, Lakewood, Colorado
  - Furiex Research Site, Longmont, Colorado
  - Furiex Research Site, Norwalk, Connecticut
  - Furiex Research Site, Ridgefield, Connecticut
  - Furiex Research Site, Boca Raton, Florida
  - Furiex Research Site, Brandon, Florida
  - Furiex Research Site, Clearwater, Florida
  - Furiex Research Site, Cooper City, Florida
  - Furiex Research Site, Coral Springs, Florida
  - Furiex Research Site, Crystal River, Florida
  - Furiex Research Site, Doral, Florida
  - Furiex Research Site, Eustis, Florida
  - Furix Research Site, Hialeah, Florida
  - Furiex Research Site, Hialeah, Florida
  - Furiex Research Site, Inverness, Florida
  - Furiex Research Site, Jacksonville, Florida
  - Furiex Research Site, Kissimmee, Florida
  - Furiex Research Site, Maitland, Florida
  - Furiex Research Site, Melbourne, Florida
  - Furiex Research Site, Miami, Florida
  - Furiex Research Site, Miami Springs, Florida
  - Furiex Research Site, Miramar, Florida
  - Furiex Research Site, Naples, Florida
  - Furiex Research Site, New Port Richey, Florida
  - Furiex Research Site, New Smyrna Beach, Florida
  - Furiex Research Site, Orlando, Florida
  - Furiex Research Site, Ormond Beach, Florida
  - Furiex Research Site, Oviedo, Florida
  - Furiex Research Site, Palm Beach, Florida
  - Furiex Research Site, Pinellas Park, Florida
  - Furiex Research Site, Port Orange, Florida
  - Furiex Research Site, Sanford, Florida
  - Furiex Research Site, Sebastian, Florida
  - Furiex Research Site, South Miami, Florida
  - Furiex Research Site, Tampa, Florida
  - Furiex Research Site, Venice, Florida
  - Furiex Research Site, Wellington, Florida
  - Furiex Research Site, Winter Haven, Florida
  - Furiex Research Site, Winter Park, Florida
  - Furiex Research Site, Atlanta, Georgia
  - Furiex Research Site, Blue Ridge, Georgia
  - Furiex Research Site, Johns Creek, Georgia
  - Furiex Research Site, Lilburn, Georgia
  - Furiex Research Site, Oakwood, Georgia
  - Furiex Research Site, Perry, Georgia
  - Furiex Research Site, Snellville, Georgia
  - Furiex Research Site, Eagle, Idaho
  - Furiex Research Site, Addison, Illinois
  - Furiex Research Site, Chicago, Illinois
  - Furiex Research Site, Morton, Illinois
  - Furiex Research Site, Brownsburg, Indiana
  - Furiex Research Site, Evansville, Indiana
  - Furiex Research Site, Indianapolis, Indiana
  - Furiex Research Site, Clive, Iowa
  - Furiex Research Site, Davenport, Iowa
  - Furiex Research Site, Iowa City, Iowa
  - Furiex Research Site, West Des Moines, Iowa
  - Furiex Research Site, Newton, Kansas
  - Furiex Research Site, Prairie Village, Kansas
  - Furiex Research Site, Shawnee Mission, Kansas
  - Furiex Research Site, Wichita, Kansas
  - Furiex Research Site, Crestview Hills, Kentucky
  - Furiex Research Site, Hawesville, Kentucky
  - Furiex Research Site, Lexington, Kentucky
  - Furiex Research Site, Louisville, Kentucky
  - Furiex Research Site, Madisonville, Kentucky
  - Furiex Research Site, Owensboro, Kentucky
  - Furiex Research Site, Baker, Louisiana
  - Furiex Research Site, Covington, Louisiana
  - Furiex Research Site, Hammond, Louisiana
  - Furiex Research Site, Metairie, Louisiana
  - Furiex Research Site, New Orleans, Louisiana
  - Furiex Research Site, Opelousas, Louisiana
  - Furiex Research Site, Shreveport, Louisiana
  - Furiex Research Site, Bangor, Maine
  - Furiex Research Site, Annapolis, Maryland
  - Furiex Research Site, Chevy Chase, Maryland
  - Furiex Research Site, Brockton, Massachusetts
  - Furiex Research Site, Watertown, Massachusetts
  - Furiex Research Site, Ann Arbor, Michigan
  - Furiex Research Site, Southfield, Michigan
  - Furiex Research Site, Stevensville, Michigan
  - Furiex Research Site, Chaska, Minnesota
  - Furiex Research Site, Jackson, Mississippi
  - Furiex Research Site, City of Saint Peters, Missouri
  - Furiex Research Site, Jefferson City, Missouri
  - Furiex Research Site, St Louis, Missouri
  - Furiex Research Site, Billings, Montana
  - Furiex Research Site, Bellevue, Nebraska
  - Furiex Research Site, Omaha, Nebraska
  - Furiex Research Site, Las Vegas, Nevada
  - Furiex Research Site, Collingswood, New Jersey
  - Furiex Research Site, Edison, New Jersey
  - Furiex Research Site, Albuquerque, New Mexico
  - Furiex Research Site, Brooklyn, New York
  - Furiex Research Site, Endwell, New York
  - Furiex Research Site, Great Neck, New York
  - Furiex Research Site, Hartsdale, New York
  - Furiex Research Site, Kew Gardens, New York
  - Furiex Research Site, New Windsor, New York
  - Furiex Research Site, New York, New York
  - Furiex Research Site, North Massapequa, New York
  - Furiex Research Site, Poughkeepsie, New York
  - Furiex Research Site, Asheville, North Carolina
  - Furiex Research Site, Charlotte, North Carolina
  - Furiex Research Site, Durham, North Carolina
  - Furiex Research Site, Fayetteville, North Carolina
  - Furiex Research Site, Greensboro, North Carolina
  - Furiex Research Site, Hickory, North Carolina
  - Furiex Research Site, High Point, North Carolina
  - Furiex Research Site, Kinston, North Carolina
  - Furiex Research Site, Lenoir, North Carolina
  - Furiex Research Site, Raleigh, North Carolina
  - Furiex Research Site, Salisbury, North Carolina
  - Furiex Research Site, Winston-Salem, North Carolina
  - Furiex Research Site, Fargo, North Dakota
  - Furiex Research Site, Beavercreek, Ohio
  - Furiex Research Site, Berea, Ohio
  - Furiex Research Site, Centerville, Ohio
  - Furiex Research Site, Cincinnati, Ohio
  - Furiex Research Site, Columbus, Ohio
  - Furiex Research Site, Dayton, Ohio
  - Furiex Research Site, Englewood, Ohio
  - Furiex Research Site, Franklin, Ohio
  - Furiex Research Site, Marion, Ohio
  - Furiex Research Site, Miamisburg, Ohio
  - Furiex Research Site, Middleburg Heights, Ohio
  - Furiex Research Site, Wadsworth, Ohio
  - Furiex Research Site, Zanesville, Ohio
  - Furiex Research Site, Tulsa, Oklahoma
  - Furiex Research Site, Belle Vernon, Pennsylvania
  - Furiex Research Site, Jenkintown, Pennsylvania
  - Furiex Research Site, Johnstown, Pennsylvania
  - Furiex Research Site, Lansdale, Pennsylvania
  - Furiex Research Site, Philadelphia, Pennsylvania
  - Furiex Research Site, Pittsburgh, Pennsylvania
  - Furiex Research Site, Uniontown, Pennsylvania
  - Furiex Research Site, Upper Saint Clair, Pennsylvania
  - Furiex Research Site, Cumberland, Rhode Island
  - Furiex Research Site, East Providence, Rhode Island
  - Furiex Research Site, Anderson, South Carolina
  - Furiex Research Site, Charleston, South Carolina
  - Furiex Research Site, Fort Mill, South Carolina
  - Furiex Research Site, Greenville, South Carolina
  - Furiex Research Site, Greer, South Carolina
  - Furiex Research Site, Myrtle Beach, South Carolina
  - Furiex Research Site, Simpsonville, South Carolina
  - Furiex Research Site, Summerville, South Carolina
  - Furiex Research Site, Bristol, Tennessee
  - Furiex Research Site, Chattanooga, Tennessee
  - Furiex Research Site, Clarksville, Tennessee
  - Furiex Research Site, Columbia, Tennessee
  - Furiex Research Site, Franklin, Tennessee
  - Furiex Research Site, Johnson City, Tennessee
  - Furiex Research Site, Memphis, Tennessee
  - Furiex Research Site, Smyrna, Tennessee
  - Furiex Research Site, Austin, Texas
  - Furiex Research Site, Baytown, Texas
  - Furiex Research Site, Beaumont, Texas
  - Furiex Research Site, Dallas, Texas
  - Furiex Research Site, El Paso, Texas
  - Furiex Research Site, Houston, Texas
  - Furiex Research Site, Marshall, Texas
  - Furiex Research Site, Plano, Texas
  - Furiex Research Site, San Antonio, Texas
  - Furiex Research Site, Sugar Land, Texas
  - Furiex Research Site, Clinton, Utah
  - Furiex Research Site, Draper, Utah
  - Furiex Research Site, Logan, Utah
  - Furiex Research Site, Ogden, Utah
  - Furiex Research Site, Salt Lake City, Utah
  - Furiex Research Site, West Jordan, Utah
  - Furiex Research Site, Lynchburg, Virginia
  - Furiex Research Site, Richmond, Virginia
  - Furiex Research Site, Williamsburg, Virginia
  - Furiex Research Site, Spokane, Washington
  - Furiex Research Site, Wenatchee, Washington
  - Furiex Research Site, Morgantown, West Virginia
  - Furiex Research Site, Wauwatosa, Wisconsin
- Canada (9):
  - Furiex Research Site, Kamloops, British Columbia
  - Furiex Research Site, Kelowna, British Columbia
  - Furiex Research Site, Winnipeg, Manitoba
  - Furiex Research Site, Bridgewater, Nova Scotia
  - Furiex Research Site, Halifax, Nova Scotia
  - Furiex Research Site, Cambridge, Ontario
  - Furiex Research Site, London, Ontario
  - Furiex Research Site, Niagara Falls, Ontario
  - Furiex Research Site, Oshawa, Ontario
- United Kingdom (16):
  - Furiex Research Site, Chesterfield, Derbyshire
  - Furiex Research Site, Blackpool, Lancashire
  - Furiex Research Site, Thornton-Cleveleys, Lancashire
  - Furiex Research Site, Burbage, Leicestershire
  - Furiex Research Site, Royal Leamington Spa, Warwickshire
  - Furiex Research Site, Chippenham, Wiltshire
  - Furiex Research Site, Bath
  - Furiex Research Site, Coventry
  - Furiex Research Site, Dorking
  - Furiex Research Site, Haxey
  - Furiex Research Site, London
  - Furiex Research Site, Shrewsbury
  - Furiex Research Site, Southampton
  - Furiex Research Site, Strensall
  - Furiex Research Site, Thornton
  - Furiex Research Site, Torpoint

REFERENCES:
- [Derived] Fant RV, Henningfield JE, Cash BD, Dove LS, Covington PS. Eluxadoline Demonstrates a Lack of Abuse Potential in Phase 2 and 3 Studies of Patients With Irritable Bowel Syndrome With Diarrhea. Clin Gastroenterol Hepatol. 2017 Jul;15(7):1021-1029.e6. doi: 10.1016/j.cgh.2017.01.026. Epub 2017 Feb 3. PMID 28167156
- [Derived] Lembo AJ, Lacy BE, Zuckerman MJ, Schey R, Dove LS, Andrae DA, Davenport JM, McIntyre G, Lopez R, Turner L, Covington PS. Eluxadoline for Irritable Bowel Syndrome with Diarrhea. N Engl J Med. 2016 Jan 21;374(3):242-53. doi: 10.1056/NEJMoa1505180. PMID 26789872

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Started | 429 | 426 | 427
Attended Week 12 Visit | 341 | 330 | 342
Attended Week 26 Visit | 289 | 291 | 290
Completed | 257 | 257 | 269
Not Completed | 172 | 169 | 158
Not completed — Voluntarily withdrew | 94 | 79 | 96
Not completed — Adverse Event | 36 | 45 | 16
Not completed — Lost to Follow-up | 25 | 23 | 16
Not completed — Physician decision: other | 11 | 14 | 16
Not completed — Physician decision: lack of efficacy | 2 | 3 | 7
Not completed — Protocol Violation | 3 | 4 | 4
Not completed — Sponsor decision | 1 | 0 | 3
Not completed — Randomized and never dispensed drug | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled Set included 1282 participants who were randomized or received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo | Total
Number analyzed (Participants) | 429 | 426 | 427 | 1282
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (13.18) | 44.4 (13.91) | 45.8 (14.10) | 44.9 (13.74)
Age, Customized [Count of Participants; unit: Participants]
  18-40 years | 173 | 166 | 159 | 498
  41-64 years | 227 | 225 | 217 | 669
  ≥65 years | 29 | 35 | 51 | 115
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 278 | 283 | 277 | 838
  Male | 151 | 143 | 150 | 444
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 374 | 368 | 370 | 1112
  Black | 46 | 48 | 46 | 140
  Asian | 3 | 3 | 4 | 10
  American Indian or Alaska Native | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Other | 5 | 4 | 6 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 119 | 117 | 125 | 361
  Not Hispanic or Latino | 310 | 309 | 302 | 921
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: The number analyzed indicates number of participants analyzed for this baseline characteristics.
  kg/m^2
    number analyzed (Participants) | 428 | 424 | 425 | 1277
    (all) | 30.70 (7.421) | 31.22 (7.858) | 30.63 (7.253) | 30.85 (7.513)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Composite Responders Based on Improvements From Baseline in Daily Worst Abdominal Pain And Daily Stool Consistency Scores
Description: Composite responders were defined as a participant who met the daily response criteria for at least 50% of the days with diary entries during the interval of interest. A participant must had met both of the following criteria on a given day to be a daily responder: 1) Daily pain response: worst abdominal pain scores in the past 24 hours improved by ≥30% compared to baseline (average of daily worst abdominal pain the week prior to randomization). 2) Daily stool consistency response: Bristol Stool Scale (BSS) score <5 (ie, score of 1, 2, 3, or 4) or the absence of a bowel movement if accompanied by ≥30% improvement in worst abdominal pain compared to baseline pain. Bristol stool scale was defined as 7-point Scale in which a score of 1 = separate hard lumps, 2 = sausage shaped but lumpy, 3 = sausage-like with cracks on the surface, 4 = sausage-like but smooth and soft, 5 = soft blobs with clear cut edges, 6 = fluffy pieces with ragged edges, and 7 = watery with no solid pieces.
Time Frame: Up to 12 Weeks
Population: Intent to Treat (ITT) analysis set included all participants who were randomized into a treatment group and presents data for participants according to their randomization assignment.
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 427 | 426 | 427
percentage of participants | 23.9 | 25.1 | 17.1
Statistical Analysis 1: Comparison: Eluxadoline 75 mg vs Placebo; The family-wise error rate was controlled by Bonferroni adjustment for each active dose versus placebo; Test type: Superiority; p = 0.014, Chi-square test statistic — Significance level of 0.025
Statistical Analysis 2: Comparison: Eluxadoline 100 mg vs Placebo; The family-wise error rate was controlled by Bonferroni adjustment for each active dose versus placebo; Test type: Superiority; p = 0.004, Chi-square test statistic — Significance level of 0.025

2. Secondary Outcome: Percentage of Participants Who Were Composite Responders Based on Improvements From Baseline in Daily Worst Abdominal Pain And Daily Stool Consistency Scores
Description: as for outcome 1
Time Frame: Up to 26 Weeks
Population: ITT analysis set included all participants who were randomized into a treatment group and presents data for participants according to their randomization assignment.
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 427 | 426 | 427
percentage of participants | 23.4 | 29.3 | 19.0
Statistical Analysis 1: Comparison: Eluxadoline 75 mg vs Placebo; The family-wise error rate was controlled by Bonferroni adjustment for each active dose versus placebo; Test type: Superiority; p = 0.112, Chi-square test statistic — Significance level of 0.025
Statistical Analysis 2: Comparison: Eluxadoline 100 mg vs Placebo; The family-wise error rate was controlled by Bonferroni adjustment for each active dose versus placebo; Test type: Superiority; p < 0.001, Chi-square test statistic — Significance level of 0.025

3. Secondary Outcome: Percentage of Participants Who Were Pain Responders In Daily Worst Abdominal Pain Scores by Intervals
Description: Pain responders were defined as participants who met the daily pain response criteria (ie, the worst abdominal pain score in the past 24 hours improved by ≥30% compared to baseline) for at least 50% of days with diary entries during each interval. A participant must have had a minimum of 20 days of diary entries over any 4-week interval, a minimum of 60 days of diary entries over the 12-week interval, and a minimum of 110 days of diary entries over the 26-week interval to be a responder.
Time Frame: 12-week interval (Weeks 1-12), 26-week interval (Weeks 1-26), and 4-week interval (Weeks 1-4, 5-8, 9-12, 13-16, 17-20, and 21-24)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 427 | 426 | 427
percentage of participants
  Responders during Weeks 1-12 | 42.4 | 43.2 | 39.6
  Responders during Weeks 1-26 | 45.2 | 46.5 | 43.3
  Responders during Weeks 1-4 | 40.5 | 44.4 | 37.5
  Responders during Weeks 5-8 | 44.5 | 47.2 | 45.4
  Responders during Weeks 9-12 | 44.5 | 45.8 | 43.8
  Responders during Weeks 13-16 | 44.3 | 44.1 | 45.4
  Responders during Weeks 17-20 | 44.7 | 43.2 | 41.5
  Responders during Weeks 21-24 | 44.7 | 42.0 | 38.4

4. Secondary Outcome: Percentage of Participants Who Were Responders In Daily Stool Consistency Scores by Intervals
Description: Stool consistency responders: participants who met daily stool consistency response criterion (ie,score of 1, 2, 3, or 4 or absence of bowel movement if accompanied by ≥30% improvement in worst abdominal pain compared to baseline pain) for at least 50% of days with diary entries during each interval. BSS was defined as 7-point Scale in which score of 1= separate hard lumps, 2= sausage shaped but lumpy, 3= sausage-like with cracks on the surface, 4= sausage-like but smooth and soft, 5= soft blobs with clear cut edges, 6= fluffy pieces with ragged edges, and 7= watery with no solid pieces. A participant must have had a minimum of 20 days of diary entries over any 4-week interval, a minimum of 60 days of diary entries over 12-week interval, and a minimum of 110 days of diary entries over 26-week interval to be a responder.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 427 | 426 | 427
percentage of participants
  Responders during Weeks 1-12 | 30.0 | 34.3 | 22.0
  Responders during Weeks 1-26 | 28.1 | 34.0 | 24.1
  Responders during Weeks 1-4 | 28.8 | 31.5 | 19.0
  Responders during Weeks 5-8 | 31.1 | 35.2 | 24.1
  Responders during Weeks 9-12 | 29.0 | 35.2 | 24.6
  Responders during Weeks 13-16 | 27.6 | 32.9 | 24.4
  Responders during Weeks 17-20 | 31.9 | 31.5 | 23.7
  Responders during Weeks 21-24 | 30.2 | 30.3 | 24.4

5. Secondary Outcome: Percentage of Participants Who Were Responders In Irritable Bowel Syndrome, Diarrhea Predominant (IBS-d) Global Symptom Scale by Intervals
Description: IBS-d global symptom responders were defined as those participants who met the daily IBS-d global symptom response criteria (ie, IBS-d global symptom score of 0 [none] or 1 [mild]; or a daily IBS-d global symptom score improved by ≥2.0 compared to the baseline average) for at least 50% of days with diary entries during each interval. IBS-d Global Symptom Scale was a 5 point scale, score ranging from 0 to 4. 0= no symptoms, 1= mild symptoms, 2= moderate symptoms, 3= severe symptoms and 4 = very severe symptoms. A participant must have had a minimum of 20 days of diary entries over any 4-week interval, a minimum of 60 days of diary entries over the 12-week interval, and a minimum of 110 days of diary entries over the 26-week interval to be a responder.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 427 | 426 | 427
percentage of participants
  Responders during Weeks 1-12 | 35.1 | 34.7 | 28.8
  Responders during Weeks 1-26 | 36.3 | 37.1 | 32.3
  Responders during Weeks 1-4 | 32.6 | 31.9 | 26.9
  Responders during Weeks 5-8 | 37.0 | 38.7 | 32.8
  Responders during Weeks 9-12 | 35.6 | 36.6 | 34.0
  Responders during Weeks 13-16 | 35.8 | 35.9 | 35.4
  Responders during Weeks 17-20 | 37.5 | 36.4 | 33.3
  Responders during Weeks 21-24 | 36.8 | 35.2 | 29.5

6. Secondary Outcome: Percentage of Participants Who Were Responders to the Irritable Bowel Syndrome Quality of Life Measure (IBS-QoL) Scale
Description: IBS-QoL responders were defined as participants who achieved at least a 14-point improvement in IBS-QoL total score from baseline to the applicable visit. The IBS-QoL consists of 34 items each with a 5-point response scale, where 1 generally represents better responses on items and 5 represents worse responses. The individual responses to the answered items were summed and standardized for a total score and then transformed to a 0- to 100-point (0= worst; 100=better) scale for ease of interpretation.
Time Frame: Weeks 4, 8, 12, 18, 26, 36, 44, and 52 (End of Treatment [EOT])
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 427 | 426 | 427
percentage of participants
  Responders at Week 4 | 42.6 | 44.1 | 37.0
  Responders at Week 8 | 43.8 | 49.8 | 41.7
  Responders at Week 12 | 44.3 | 48.1 | 44.0
  Responders at Week 18 | 44.5 | 45.1 | 43.3
  Responders at Week 26 | 45.4 | 45.1 | 40.0
  Responders at Week 36 | 41.0 | 43.2 | 39.6
  Responders at Week 44 | 39.6 | 40.1 | 37.5
  Responders at Week 52/EOT | 49.4 | 54.9 | 47.8

7. Secondary Outcome: Percentage of Participants With Irritable Bowel Syndrome - Adequate Relief (IBS-AR) Scale
Description: Adequate relief of IBS symptoms was assessed once weekly by participants answering the IBS-AR item in the electronic diary. IBS-AR responders were defined as participants with a weekly response of "Yes" to adequate relief of their IBS symptoms for at least 50% of the total weeks during the interval. A participant must have had a positive response on ≥6 weeks for the 12-week interval and ≥13 weeks for the 26-week interval, regardless of diary compliance, to be a responder.
Time Frame: 12-week interval (Weeks 1-12) and 26-week interval (Weeks 1-26)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 427 | 426 | 427
percentage of participants
  Responders during Weeks 1-12 | 52.9 | 54.2 | 43.8
  Responders during Weeks 1-26 | 45.7 | 49.5 | 40.0

8. Secondary Outcome: Change From Baseline in Daily Abdominal Discomfort Scores
Description: Symptoms of abdominal discomfort were recorded on a 0 to 10 scale, where 0 corresponded to no discomfort and 10 corresponded to worst imaginable discomfort. A negative change from Baseline indicates the discomfort decreased.
Time Frame: Baseline, Weeks 4, 12 and 26
Population: Intent to Treat (ITT) analysis set included all participants who were randomized into a treatment group and presents data for participants according to their randomization assignment. Here, number analyzed is the participants who were evaluable at specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 427 | 426 | 427
score on a scale
  Change at Week 4: number analyzed (Participants) | 392 | 381 | 401
  Change at Week 4 | -2.24 (2.204) | -2.41 (2.326) | -2.01 (2.156)
  Change at Week 12: number analyzed (Participants) | 338 | 335 | 335
  Change at Week 12 | -2.75 (2.534) | -2.97 (2.526) | -2.61 (2.444)
  Change at Week 26: number analyzed (Participants) | 264 | 262 | 264
  Change at Week 26 | -3.27 (2.578) | -3.52 (2.543) | -3.00 (2.579)

9. Secondary Outcome: Change From Baseline in Daily Abdominal Bloating Scores
Description: Symptoms of abdominal bloating were recorded on a 0 to 10 scale, where 0 corresponded to no bloating and 10 corresponded to worst imaginable bloating. A negative change from Baseline indicates the bloating decreased.
Time Frame: Baseline, Weeks 4, 12 and 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 427 | 426 | 427
score on a scale
  Change at Week 4: number analyzed (Participants) | 330 | 318 | 329
  Change at Week 4 | -1.84 (2.303) | -2.03 (2.333) | -1.72 (2.303)
  Change at Week 12: number analyzed (Participants) | 277 | 272 | 274
  Change at Week 12 | -2.42 (2.616) | -2.49 (2.533) | -2.16 (2.544)
  Change at Week 26: number analyzed (Participants) | 209 | 210 | 210
  Change at Week 26 | -2.76 (2.823) | -2.94 (2.576) | -2.47 (2.562)

10. Secondary Outcome: Number of Bowel Movements Per Day
Description: Participants recorded the number of bowel movements over 24 hours daily throughout the treatment.
Time Frame: Weeks 4, 12 and 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: bowel movements per day
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 427 | 426 | 427
bowel movements per day
  Week 4: number analyzed (Participants) | 392 | 381 | 401
  Week 4 | 3.20 (2.090) | 3.20 (2.236) | 3.72 (2.100)
  Week 12: number analyzed (Participants) | 338 | 335 | 335
  Week 12 | 3.12 (2.143) | 3.09 (2.318) | 3.44 (1.987)
  Week 26: number analyzed (Participants) | 264 | 262 | 264
  Week 26 | 2.83 (2.158) | 2.79 (2.270) | 3.12 (1.831)

11. Secondary Outcome: Number of Bowel Incontinence Episodes
Description: Participants recorded the number of incontinence episodes over 24 hours daily throughout the treatment.
Time Frame: Weeks 4, 12 and 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: incontinence episodes
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 427 | 426 | 427
incontinence episodes
  Week 4: number analyzed (Participants) | 392 | 381 | 401
  Week 4 | 0.74 (1.603) | 0.72 (1.534) | 0.93 (2.140)
  Week 12: number analyzed (Participants) | 338 | 335 | 335
  Week 12 | 0.63 (1.542) | 0.71 (1.663) | 0.94 (3.612)
  Week 26: number analyzed (Participants) | 264 | 262 | 264
  Week 26 | 0.46 (1.298) | 0.58 (1.358) | 0.69 (1.500)

12. Secondary Outcome: Number of Bowel Incontinence Free Days
Description: An incontinence free day was one where the participant reports zero incontinence episodes. The number of incontinence free days for a participant was assessed each week based on the number of reported days.
Time Frame: Weeks 4, 12 and 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 427 | 426 | 427
days
  Week 4: number analyzed (Participants) | 392 | 381 | 401
  Week 4 | 4.83 (2.745) | 4.95 (2.618) | 4.63 (2.741)
  Week 12: number analyzed (Participants) | 338 | 335 | 335
  Week 12 | 4.96 (2.672) | 4.79 (2.671) | 4.64 (2.704)
  Week 26: number analyzed (Participants) | 264 | 262 | 264
  Week 26 | 4.39 (2.465) | 4.35 (2.449) | 4.00 (2.539)

13. Secondary Outcome: Number of Urgency Episodes Per Day
Description: Participants recorded the number of urgency episodes over 24 hours daily throughout the treatment.
Time Frame: Weeks 4, 12 and 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: episodes per day
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 427 | 426 | 427
episodes per day
  Week 4: number analyzed (Participants) | 392 | 381 | 401
  Week 4 | 1.75 (1.840) | 1.74 (1.879) | 2.19 (2.082)
  Week 12: number analyzed (Participants) | 338 | 335 | 335
  Week 12 | 1.55 (1.777) | 1.60 (1.995) | 1.81 (1.883)
  Week 26: number analyzed (Participants) | 264 | 262 | 264
  Week 26 | 1.25 (1.773) | 1.45 (2.113) | 1.55 (1.853)

14. Secondary Outcome: IBS-QoL Total Scores
Description: The IBS-QoL consists of 34 items each with a 5-point response scale, where 1 generally represents better responses on items and 5 represents worse responses. The individual responses to the answered items were summed and standardized for a total score and then transformed to a 0- to 100- point scale (0=worst; 100=better) for ease of interpretation.
Time Frame: Weeks 4, 8, 12, 18, 26, 36, 44, and 52 (EOT)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 427 | 426 | 427
score on a scale
  Responders at Week 4: number analyzed (Participants) | 384 | 371 | 392
  Responders at Week 4 | 62.37 (23.747) | 64.34 (24.049) | 57.13 (24.318)
  Responders at Week 8: number analyzed (Participants) | 354 | 354 | 360
  Responders at Week 8 | 66.22 (23.919) | 67.73 (23.421) | 59.46 (24.323)
  Responders at Week 12: number analyzed (Participants) | 339 | 330 | 342
  Responders at Week 12 | 66.80 (24.131) | 68.93 (23.938) | 61.72 (25.545)
  Responders at Week 18: number analyzed (Participants) | 315 | 312 | 315
  Responders at Week 18 | 68.75 (23.902) | 70.05 (23.662) | 63.60 (24.618)
  Responders at Week 26: number analyzed (Participants) | 288 | 291 | 290
  Responders at Week 26 | 70.74 (23.312) | 71.34 (23.106) | 64.83 (24.380)
  Responders at Week 36: number analyzed (Participants) | 277 | 272 | 278
  Responders at Week 36 | 70.53 (23.043) | 72.37 (23.246) | 66.47 (24.034)
  Responders at Week 44: number analyzed (Participants) | 267 | 261 | 271
  Responders at Week 44 | 70.30 (24.408) | 72.15 (24.398) | 65.59 (25.045)
  Responders at Week 52/EOT: number analyzed (Participants) | 351 | 353 | 362
  Responders at Week 52/EOT | 68.85 (24.754) | 71.02 (24.294) | 63.93 (26.359)

15. Secondary Outcome: Change From Baseline in IBS-QoL Total Scores
Description: The IBS-QoL consists of 34 items each with a 5-point response scale, where 1 generally represents better responses on items and 5 represents worse responses. The individual responses to the answered items were summed and standardized for a total score and then transformed to a 0- to 100- point scale (0=worst; 100=better) for ease of interpretation. A positive change from Baseline indicates that quality of life improved.
Time Frame: Baseline, Weeks 4, 8, 12, 18, 26, 36, 44, and 52/EOT
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 427 | 426 | 427
score on a scale
  Change at Week 4: number analyzed (Participants) | 382 | 371 | 392
  Change at Week 4 | 16.49 (20.693) | 17.86 (20.191) | 13.25 (18.475)
  Change at Week 8: number analyzed (Participants) | 353 | 354 | 360
  Change at Week 8 | 19.88 (21.855) | 21.08 (21.347) | 15.76 (19.398)
  Change at Week 12: number analyzed (Participants) | 337 | 330 | 342
  Change at Week 12 | 20.26 (23.412) | 22.76 (22.592) | 17.76 (21.523)
  Change at Week 18: number analyzed (Participants) | 313 | 312 | 315
  Change at Week 18 | 23.09 (23.846) | 24.18 (23.025) | 19.80 (22.368)
  Change at Week 26: number analyzed (Participants) | 288 | 291 | 290
  Change at Week 26 | 25.28 (23.679) | 25.80 (23.998) | 20.62 (22.306)
  Change at Week 36: number analyzed (Participants) | 277 | 272 | 278
  Change at Week 36 | 25.37 (24.603) | 27.18 (24.201) | 22.64 (23.414)
  Change at Week 44: number analyzed (Participants) | 267 | 261 | 271
  Change at Week 44 | 25.13 (24.948) | 26.64 (25.017) | 21.77 (23.977)
  Change at Week 52/EOT: number analyzed (Participants) | 349 | 353 | 362
  Change at Week 52/EOT | 23.30 (23.959) | 25.86 (23.854) | 20.66 (23.956)

ADVERSE EVENTS:
Time Frame: Up to 54 weeks
Description: The Safety Analysis Set included enrolled participants who received at least one dose of study drug and presents data according to the actual treatment received. A total of 53 participants were randomized to the Eluxadoline 75 mg arm but received Eluxadoline 100 mg due to site misallocations, these participants were included in Eluxadoline 100 mg arm. Therefore, the number of participants in the Eluxadoline 100 mg arm were more than the number of participants who were randomized to this arm.
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/428 | 0/479 | 0/427
Serious Adverse Events (participants affected / at risk) | 25/428 | 27/479 | 16/427
Other Adverse Events (participants affected / at risk) | 84/428 | 89/479 | 47/427
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eluxadoline 75 mg (N=428) | Eluxadoline 100 mg (N=479) | Placebo (N=427)
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum intestinal hemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Primary progressive multiple sclerosis (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hematoma (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural hematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 1
Conversion disorder (Psychiatric disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Papilloedema (Eye disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Abortion spontaneousa (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eluxadoline 75 mg (N=428) | Eluxadoline 100 mg (N=479) | Placebo (N=427)
Constipation (Gastrointestinal disorders) | 27 | 44 | 12
Nausea (Gastrointestinal disorders) | 34 | 31 | 19
Vomiting (Gastrointestinal disorders) | 22 | 19 | 7
Upper respiratory tract infection (Infections and infestations) | 14 | 25 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will work with the Investigators to determine how any manuscript or publication in a scientific journal is written and edited, the number and order of authors, the publication to which it will be submitted, and other related issues. The sponsor has final approval authority over all such issues. Data are the property of the sponsor and cannot be published without prior authorization from the sponsor, but data and publication thereof will not be unduly withheld.